CLINICAL TRIAL: NCT01605682
Title: Multi Dose Effects of a Berry Extract Upon Mood, Attention and Memory in Healthy Young Adults.
Brief Title: Multi Dose Effects of a Berry Extract Upon Moodand Cognition in Healthy Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Collaborators: The New Zealand Institute of Plant and Food Research Ltd. (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: 28AI2
Record Dates: First submitted 2012-05-17; First posted 2012-05-25 (Estimated); Last update posted 2012-05-25 (Estimated); Status verified 2012-05

CONDITIONS: Healthy
Keywords: effect of different berry doses on mood and cognition; adults

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Berry extract 125 (Experimental): Fresh berry extract containing 125mg of polyphenols
  Interventions: Dietary Supplement: Fresh berry extract.
- Berry extract 250 (Experimental): Fresh berry extract containing 250mg of polyphenols
  Interventions: Dietary Supplement: Fresh berry extract.
- Berry extract 500 (Experimental): Fresh berry extract containing 500mg of polyphenols
  Interventions: Dietary Supplement: Fresh berry extract.
- Placebo (Placebo Comparator): Berry flavoured juice containing no polyphenols
  Interventions: Dietary Supplement: Fresh berry extract.

INTERVENTIONS:
Dietary Supplement: Fresh berry extract. — Fresh berry extract containing 500mg, 250mg, 125mg per 60 kilos of body weight. Or placebo.

SUMMARY:
Berry fruits are widely recognised as natural functional food products. They contain several different phytochemicals which have potential to modulate human health and wellbeing. There is however some debate regarding the mechanisms driving their health promoting properties.

Despite the wide health promoting properties of fruit extracts reported in the literature, considerable interest over the past decade has primarily been focused on their roles in reducing risk factors associated with cancer and heart disease. Consequently, there remains a paucity of actual scientific information on their role in modulating brain functions, such as mood, learning and memory, any decrements of which have very negative impacts on the quality of life.

A prior study carried out as the first study of my PhD, attempted to bridge this gap in knowledge and found promising results after acutely supplementing participants with a fruit based drink. The findings showed that there was an increased vigilance on attention related psychometric tasks and an increased feeling of calmness. The investigators have hypothesised that these cognitive enhancing effects are due to the monoamine oxidase (MAO) inhibiting effect of the fruit drink, our ex vivo findings support this with a 96% reduction in MAO-B activity.

The aims of the current study are threefold: to extend the findings of my previous investigation by extending the tasks explored; to ascertain if the positive results of the first study are dose dependent; and to investigate whether a lower dose can facilitate greater changes in behaviour.

DETAILED DESCRIPTION:
The project will investigate the acute effects on human cognitive behaviour and mood of a single consumption of 3 fruit drinks versus a placebo. Drinks will be matched for volume, taste, appearance and sugars but will differ in the amount of total polyphenols. The 3 active treatment drinks contain a natural berry fruit grown in New Zealand by Plant and Food Research from commercial cultivars.

The study will follow a double-blind, counterbalanced, placebo controlled, repeated measures, crossover design with 36 healthy participants aged between 18 and 35 completing four study day sessions as well as one training/screening visit (five visits in total). On one occasion participants will receive a placebo, on another fruit drink 1, on another fruit drink 2 and on another fruit drink 3. Study days will be spaced one week apart to accommodate a wash out period. Fruit drinks will be made to include 500mg, 250mg or 125mg of polyphenols/60kg of body weight. Sucralose (artificial sweetener) will be added to make the drinks palatable. Participants will be screened for any intolerance or allergies to the drinks during the training/screening session . Trait anxiety will also be assessed during the screening visit using the State-Trait Anxiety inventory (STAI - Spielberger, 1966).

Psychometric tasks and mood scales will be delivered using the Computerised Mental Performance Assessment System (COMPASS), a purpose designed software application for the flexible delivery of randomly generated parallel versions of standard and novel cognitive assessment tasks that has previously been shown to be sensitive to nutritional interventions. .

Baseline cognitive testing will involve the dual task, Digit vigilance, Digit vigilance fast, Visual analogue scales, 3-back, corsi blocks, simple reaction time, telephone number task, word recognition, word recall, Bond-Lader mood scales and the state anxiety questionnaire (STAI).

Baseline On all 3 testing days participants will arrive at the lab in the morning (8:00 am), after an overnight fast, and firstly give a 10 mL venous blood sample taken by a trained phlebotomist. Participants will then complete one repetition of the COMPASS computerised cognitive assessment battery (baseline). Participants will then be orally supplemented with treatment in the form of a single serve juice drink (200ml per 60kg weight).

Post Supplementation 60 minutes after supplementation, the first post dose state anxiety questionnaire will be completed. Participants will then complete the first post dose COMPASS assessment. After completion of the assessment participants will immediately give a second 10 ml venous blood sample. Participants will then have a 20 minute break before completing the second post dose COMPASS assessment and complete a final post dose state anxiety questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* aged between 18-35 years old,
* non smokers,
* bmi < 30kg/m2

Exclusion Criteria:

* smoker,
* pregnant,
* currently taking recreational over the counter/prescription medication (excluding the contraceptive pill) and/or dietary/herbal supplements.
* food allergies or sensitivities that are relevant to the study,
* learning difficulties,
* ADHD,
* dyslexia,
* migraines or
* any gastric problems

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2011-07; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Change in cognition | baseline, 1 hour post dose and 2 hours 30mins post dose.
Change in mood | Baseline, 1 hour post dose and 2 hours 30mins post dose.
Change in Monoamine Oxidase-B activity | baseline and 2 hours post dose

SECONDARY OUTCOMES:
Change in prolactin | baseline and 2 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Anthony w Watson, Principal Investigator — Northumbria University
Locations (1):
- The Brain Performance and Nutrition Research Center, Newcastle upon Tyne, United Kingdom